CLINICAL TRIAL: NCT06571838
Title: DAISY: Diagnostic AI System for Robotic and Automated Triage and Assessment
Brief Title: DAISY- Diagnostic AI System for Robotic and Automated Triage and Assessment
Acronym: DAISY
Status: Recruiting | Type: Observational
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of York (Other)
Responsible Party: Sponsor
Other Study IDs: 343550
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DAISY system — DAISY is a The humanoid robot with an ipad and attached peripheral devices capable of taking blood pressure and temperature

SUMMARY:
This study aims to introduce an automated triaging system called DAISY into the Emergency Department (ED) to give patients the opportunity to self-direct their initial consultation. This is a new system in development, with a robot like the image at the top of this sheet, a touchscreen that will ask patients a number of questions about their current health (as a Triage nurse or doctor in the Emergency Department may do) but also with some attached devices (like a blood pressure monitor and thermometer) that patients can use to help DAISY assess patients' current health.

This study aims to demonstrate how patients can interact with the automated system to produce a report that is useful for the doctors and nurses in the ED. The study will examine the duration and timeliness of the automated assessment to see if it frees up staff time and determine how patients find the experience of using the DAISY system.

DETAILED DESCRIPTION:
The number of patients arriving at Emergency Departments (EDs) in England increased by 21% between 2010 and 2019. Combined with international healthcare staff shortages which have been an ongoing concern for over three decades, this has resulted in overcrowded EDs and long patient waits. Over 20,000 patients waited more than 12 hours for treatment in EDs in England in December 2021. As such, solutions must be explored to alleviate the strain on medical professionals and systems so that they can optimise their time,and increase the throughput in EDs for the benefit of patients.

The use of digital technology to collect, organise and perform initial analysis of patients without the need to interact with healthcare staff, theoretically frees staff from data collection, reducing waiting times and the door-to-treatment times. DAISY is a proposed humanoid Robot that uses digital technology to perform these 'front-door' functions.

The trial participants will be patients who self-present to the Emergency Department with acute clinical needs. The study is unblinded and adult ED users are invited to participate in the use of an automated triage process while they await the regular human triage personnel. Potential participants may be primarily identified by the reception staff after which they undergo an initial screening by a member of the investigating team who consents the patient for the study according to the protocol specifications. The participants, thereafter interact with DAISY to complete a consultation after which an anonymised report is generated as the initial Case Report Form (CRF). The participant returns to their original position in the traditional triage queue without an advantage or disadvantage in the 'time-to-see' a clinician. Their return signifies the end of their active participation in the trial.

Participants are expected to spend less than 30 minutes for the automated consultation. They may choose to discontinue their engagement with the study at any point during the process. Participants who do not complete the process will be included in the final data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* Aged 18 years or above
* Able and willing to comply with all study requirements
* Able to engage or operate the automated system, either unaided or with help from own carers

Exclusion Criteria:

* Less than 18 years of age
* Decreased consciousness and/or affect
* In need of urgent transfer to the resuscitation area
* Deemed unsuitable or too unwell by the recruiting investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years of age attending the Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 30 minutes
  Patient feedback scores

SECONDARY OUTCOMES:
Duration | 30 minutes
  Time taken for the consultation process
Engagement | 30 minutes
  Patient satisfaction scores with the automated process
Concordance | 30 minutes
  Level of concordance between DAISY report and human generated report

CONTACTS AND LOCATIONS:
Locations (1):
- York & Scarborough Teaching Hospitals NHS Foundation Trust, York, N. Yorks, United Kingdom

IPD SHARING:
Plan to Share IPD: No